# Clinical Investigation Plan

# **CP363**

Clinical Investigation Exploring Two Ostomy Product Prototypes

November 2023-March 2024

Master

ClinicalTrials.gov ID: NCT06237686

Approval date of version 2.0: 2023/12/19

### **CHANGE LOG**

| VERSION<br>NUMBER | ISSUED BY<br>(INITIALS) | COMMENTS (MAJOR CHANGES SINCE LAST REVISION) |
|---|---|---|
| 1.0 | | First approved version |
| 2.0 | | |

This confidential document is the property of Coloplast A/S. No unpublished information contained herein may be disclosed without written approval of Coloplast A/S.

### SYNOPSIS OF THE CLINICAL INVESTIGATION

#### Title

### Clinical Investigation Exploring Two Ostomy Product Prototypes

#### Test products

Two ostomy product prototypes (Test product A and B) will be tested in this investigation.

#### Intended use

The test products are intended to be used in the same manner as a CE-marked ostomy product.

### Objective(s)

### Primary objective

The primary objective is to investigate Test product A and B's ability to swell around the stoma.

### Secondary objective

The secondary objective is to investigate the peristomal skin condition after wearing Test products A and B for 4 hours.

# Design of the investigation

The clinical investigation is a non-comparative, one-sequence, open-labelled, single-centre study.

### Expected duration of the clinical investigation

All subjects will test both Test product A and B, with a minimum of 7 days apart. In total, each subject will be enrolled in the investigation for 8 days +3 days.

### Primary endpoint and secondary endpoint(s)

### Primary endpoint

The Test product formulation's ability to swell at the end of each test period (assessed by photos and video by qualitative evaluation).

### Secondary endpoint

The change in pain, itching and burning (PIB) score (0-10) based on Peristomal Skin Health (The Ostomy Skin Tool 2.0) from before to after end use of the Test products.



Adverse events

## Population/subjects

As this is an exploratory investigation with a qualitative primary outcome no formal sample size is calculated but it is evaluated that 10 subjects with an ileostomy (liquid output) will be adequate to investigate the Test product A and B's ability to swell around the stoma.

| Inclu | Inclusion criteria | | Exclusion criteria |
|---|---|---|---|
| To be included in this investigation the subject must answer yes to the following inclusion criteria's: | | To be included in this investigation the subject must answer no to the following exclusion criteria's: | |
| 1. | Has given written informed consent | 1. | Is currently receiving or have within the past 60 days received radio- and/or chemotherapy (Low doses radio- and/or chemotherapy (Assessed by Principal Investigator) is allowed. for indications other than cancer) |
| 2. | Is at least 18 years of age and has full legal capacity | 2. | Is currently receiving or have within the past 30 days received topical steroid treatment in the peristomal skin area, e.g. lotion or spray or systemic steroid (tablet/injection) treatment |
| 3. | Has had an ileostomy for more than 3 months | 3. | Is pregnant or breastfeeding |
| 4. | Has suitable peristomal skin area (assessed by investigator) | 4. | Has dermatological problems in the peristomal area (assessed by investigator) |
| 5. | Is currently using flat SenSura Mio 1-piece or 2-piece | 5. | Participates in other clinical investigations. Exception: Participation in other Coloplast sponsored clinical investigations is accepted under the circumstances that the subject has paused the activities in the investigation and are otherwise complying with the inclusion and exclusion criteria of this protocol |
| 6. | Has used flat SenSura Mio 1-piece or 2-piece for at least 14 days | 6. | Has any known allergies towards ingredients in the investigational device |
| 7. | Has a stoma size less than 45mm in diameter | | |

# LIST OF ABBREBIATIONS

| ABBREVIATION | WRITTEN OUT | EXPLANATION |
|---|---|---|
| ADE | Adverse Device Effect | See section 18.2 |
| AE | Adverse Event | See section 18.1 |
| ASADE | Anticipated Serious Adverse Device Effect | See section 18.4.2 |
| CIP | Clinical Investigation Plan | |
| CRF | Case Report Form (paper or electronic) | Questionnaire to be used for data collection |
| СМ | Clinical Manager | |
| DQF | Data Query Forms | A DQF is a query specifically used in clinical research. The DQF is the primary data query tool from the sponsor to clarify discrepancies and ask the investigator for clarification. The DQF is part of the data validation process in a clinical investigation. |
| DD | Device deficiency | |
| EC | Ethics Committee | |
| IB | Investigator's Brochure | Compilation of the current clinical and non-clinical information on<br>the investigational medical device(s,) relevant to the clinical in-<br>vestigation. |
| IFU | Instruction For Use | |
| ITT | Intention to Treat | |
| Pl | Principal Investigator | Qualified person responsible for conducting the clinical investigation at an investigation site. If the clinical investigation is conducted by a team of individuals at an investigation site, the PI is the responsible leader of the team. Whether this is the responsibility of an individual or an institution can depend on national regulations. |
| PP | Per Protocol | |
| SADE | Serious Adverse Device Effect | See section 18.4.1 |
| SAE | Serious Adverse Event | See section 0 |
| USADE | Unanticipated Serious Adverse Device Effect | See section 0 |

# > TABLE OF CONTENTS

| 1. | List of personnel involved in the Investigation8 |
|---|---|
| 1.1. | Sponsor representatives8 |
| 1.2. | Investigators8 |
| 2. | Rational/justification for conducting the clinical investigation8 |
| 3. | Objective(s) and hypotheses of the clinical investigation9 |
| 3.1. | Objective (s)9 |
| 3.2. | Hypotheses9 |
| 4. | Investigational device and comparator(s)9 |
| <b>4.1.</b> 4. | 1.1. Manufacturing |
| 4.2. | |
| 4.3. | ##################################### |
| 4.4. | |
| 4.5. | Handling of the investigational device10 |
| 4.6. | |
| 4.7. | |
| <b>5</b> . | Design of the clinical investigation11 |
| 5.1. | General |
| 5.2. | |
| 5.3. | ************************************** |
| 5.4. | |
| 5.5. | • |
| 5.6. | - 1 1 |
| 5.7. | |
| 5.8. | Section (Section 2) Contraction (Section 2) Contractio |
| | Total expected duration of the clinical investigation12 |
| 6. | Clinical Investigation population12 |
| 6.<br>6. | 1.1. Inclusion criteria 13 1.2. Exclusion criteria 13 1.3. Pregnancy and breastfeeding 14 1.4. Vulnerable population (If applicable) 14 |
| 6.2. | |
| 6.3. | • |
| 64 | Point of enrolment 15 |

| 6.5 | . s | Subject Identification and Confidentiality | 15 |
|---|---|---|---|
| 7. | Pro | ocedures | 16 |
| 7.1 | | Clinical investigation-related procedures | 16 |
| 7.2 | F | low-chart | 17 |
| 7.3 | | Concomitant treatment | 19 |
| 8. | Ris | sk – benefit analysis and ethical considerations | 19 |
| 8.1. | | Risk-benefit analysis of the investigational device | |
| 8.2 | R | Risk-benefit for subjects participating in the clinical investigation | 19 |
| 8.3 | R | Risk Analysis for the conduct of the clinical investigation | 20 |
| 8.4 | D | Delegation of responsibility | 20 |
| 9. | Mo | nitoring activities | 20 |
| 9.1. | S | site visits | |
| | 1.1. | | 20<br>20 |
| | 1.3. | | 20 |
| 9.2. | R | Remote monitoring | 21 |
| 9.3. | S | ource data verification | 22 |
| 10. | Sta | atistical considerations | 22 |
| 10. | 1. | Statistical design, method and analytical procedures | 22 |
| 10. | 2. | Sample size | 23 |
| 10.3 | 3. | Level of significance and power | 23 |
| 10.4 | 4. | Pass/fail criteria | 23 |
| 10. | 5. | Interim analysis | 23 |
| 10.0 | 6. | Statistical reason for termination of investigation | 23 |
| 10. | 7. | Deviation(s) from statistical design, method or analytical procedures | 23 |
| 11. | Da | ta management | 23 |
| 11. | 1. | Data collection procedure | 24 |
| 11.3 | 2. | Data retention | 25 |
| 12. | Am | nendments to the Clinical Investigation Plan | 25 |
| 13. | De | viations from the Clinical Investigation Plan | 25 |
| 14. | De | vice Accountability | 26 |
| 15. | | atement of compliance | |
| 15. | | Ethics committee and regulatory authorities | |
| 15. | 2. | Data protection | |
| 15. | 3. | Indemnity | |
| 15.4 | 4. | Financial conditions | |
| 16. | Info | ormed consent process | 27 |
| 17 | | hiect compensation | |

| 17.1. | Compensation in case of injury | 28 |
|---|---|---|
| 17.2. | Compensation for participating in the clinical investigation | 28 |
| 18. Ad | verse events, adverse device effects and device deficiencies | 28 |
| 18.1. | Adverse events | 28 |
| 18.2. | Adverse device effect | 28 |
| 18.3. | Device deficiency | 29 |
| 18.4. | Serious adverse events (SAE) | 29 |
| 18.4.1 | | 29 |
| 18.4.2 | | |
| 18.4.3 | | |
| 18.5. | Medical care of subjects | 29 |
| 18.6. | Reporting and timelines | 30 |
| 18.7. | Investigator's reporting responsibilities | 30 |
| 18.8. | Sponsors reporting responsibilities | 31 |
| 19. Su | spension or premature termination of the clinical investigation | 31 |
| 20. Cli | nical investigation report | 31 |
| | blication policy | |
| 21.1. | General | |
| 22. Su | spension/termination of the clinical investigation | |
| | ferences | |
| | pendix | |

# 1. List of personnel involved in the Investigation.

# 1.1. Sponsor representatives

| SENIOR CLINICAL MANAGER | PRINCIPAL BIOSTATISTICIAN |
|---|---|
| SENIOR DATA MANAGEMENT SPECIALIST | CLINICAL STRATEGY PROJECT MANAGER |
| SENIOR DIRECTOR OF CLINICAL OPERATIONS | MEDICAL WRITER |

### 1.2. Investigators

The CM is responsible for maintaining an updated list of all PIs, investigation sites and institutions.



In case of emergency, please contact the CM from the above list of sponsor representatives.

# 2. Rational/justification for conducting the clinical investigation

Peristomal skin complications (PSCs) are the predominant complication for people living with a stoma, which affect their quality of life negatively (1).

Especially among people living with an ileostomy or colostomy with liquid faecal effluent, the incidence of PSCs is high (2, 3), which may be ascribed to the presence of a high content of digestive proteolytic enzymes and other chemical irritants in the liquid and corrosive effluent (4-6). Some of the common clinical signs of PSCs include pain, itching, burning, discoloration, bleeding, and wounds (3).

Among the main reasons for developing PSCs are that the peristomal skin is exposed to stomal output either due to leakage of output under the baseplate and/or imperfect cutting of the hole in the baseplate, and incorrect application creating a gap between the hole in the baseplate and the stoma (2, 3, 7).

The aim of the present investigation is to explore the properties of two different ostomy product prototypes (Test products A and B) during use.

The data from this explorative investigation will be used for further optimization and development of the prototypes.

# 3. Objective(s) and hypotheses of the clinical investigation

### 3.1. Objective (s)

### Primary objective

The primary objective is to investigate Test product A and B's ability to swell around the stoma.

### Secondary objective

The secondary objective is to investigate the peristomal skin condition after wearing Test product A and B for 4 hours.

### 3.2. Hypotheses

This is an exploratory investigation and there is no formal success and/or fail criteria and no formal hypotheses applied in this investigation. It is expected that the results of this investigation will provide valuable in-sight to the further optimization and development of the Test products (prototypes).

# 4. Investigational device and comparator(s)

Two ostomy product prototypes (Test product A and B) will be tested in this investigation.

### 4.1. Description of investigational device

The Swellertech formulations of Test product A and B are characterized as followed:

Below in fig. 1 a schematic drawing of the test product is shown.



# 4.1.1. Manufacturing

Coloplast A/S

is legal manufacturer of the test products.

## 4.2. Identification and traceability of the device

The test products will be identified as CP363/A and CP363/B.

Investigational device label can be found in Investigators Brochure (8)

### 4.3. Intended use of the device in the clinical investigation

The test products are intended to be used in the same manner as a CE-marked ostomy product.

### 4.4. Intended population for the device

The population will consist of 10 subjects with an ileostomy (liquid output). To be enrolled in the investigation, subjects must comply with the Eligibility criteria's in section 6.1.

# 4.5. Handling of the investigational device

Handling of the test products do not require specific competencies other than health care professional basic training. The test products will only be handled by study personal, who will receive training in study conduct during SIV.

Further details can be found in the IB (9)

# 4.6. Total number of devices intended for the clinical investigation

Each subject is expected to use one of each Test product A and B during their participation in the investigation.

This gives:

1x10 = 10 Test product A

1x10 = 10 Test product B

Additionally, an extra buffer of 10 x each Test product will be produced.

In total, 20 of each Test product A and B needs to be released for the investigation.

# 4.7. Description of the comparator product(s)

No comparator is used is this investigation.

# 5. Design of the clinical investigation

### 5.1. General

The clinical investigation is a non-comparative, one-sequence, open-labelled, single-centre study.

All subjects will test both Test products A and B with a minimum of 7 days apart. In total, each subject will be enrolled in the investigation for 8 days +3 days.

The study will consist of:

- V0: Information visit
- V1: Inclusion of subjects, baseline registrations and Test visit 1 (Testing Test product A)
- V2: Test visit 2 (Testing Test product B) and Termination visit

V0 and V1 can be conducted on the same day.

The test period of each Test product (A and B) is set to 4 hours. The total duration of each visit (V1 and V2) is set to approximately 5 hours. Subjects will leave each test visit using only their usual stoma product.



Figure 2 Schematic view of investigation

# 5.2. Primary endpoint

The Test product formulation's ability to swell at the end of each test period (assessed by photos and video by qualitative evaluation).

### 5.3. Secondary endpoints

The change in pain, itching and burning (PIB) score (0-10) based on Peristomal Skin Health The Ostomy Skin Tool 2.0 (OLS 2.0)) from before to after end use of the Test products.

The questions of experienced PIB underneath the centre part of the baseplate from the OST 2.0 are (see Appendix 1):

- Please rate on a scale from 0-10 how itchy the skin around your stoma has been <u>at its worst</u> since you
  last changed your product (rated on a scale from 0-10, where 0 is no itch and 10 is worst possible
  peristomal skin itch).
- Please rate on a scale from 0-10 how painful the skin around your stoma has been <u>at its worst</u> since
  you last changed your product (rated on a scale from 0-10, where 0 is no pain and 10 is worst possible
  peristomal skin pain).
- Please rate on a scale from 0-10 any burning feelings from the skin around your stoma at its worst since you last changed your product (rated on a scale from 0-10, where 0 is no burning and 10 is worst possible peristomal skin burning).



Adverse events

# 5.5. Rationale for selection and measurement of endpoints

It is expected that the selected endpoints will provide valuable in-sight to the further optimization and development of the test products (prototypes).

# 5.6. Equipment

- Ruler
- Camera

### 5.7. Randomisation Procedure

Not applicable

# 5.8. Blinding

Not applicable

## 5.9. Total expected duration of the clinical investigation

The dates below are approximate, and no subjects will be enrolled before all required approvals have been obtained. If changes are required, applicable EC will be notified.

First subject enrolled (12/2023)

Last subject enrolled (02/2024)

Last subject complete (02/2024)

Final report (02/2025)

### 6. Clinical Investigation population

The population will consist of 10 subjects with an ileostomy (liquid output) enrolled at one clinical investigation site. Screening failures and subjects who withdraw or are prematurely terminated from the investigation will be replaced until 10 subjects have completed the study.

6.1. Eligibility criteria

To be included in the investigation, the subjects must comply with the selection criteria described below.

# 6.1.1. Inclusion criteria

| | To be included in this investigation the sub-<br>ject must answer yes to the following inclu-<br>sion criteria: | Justification for inclusion criteria |
|---|---|---|
| 1. | Has given written informed consent | To meet the Helsinki declaration |
| 2. | Is at least 18 years of age and has full legal capacity | To meet the Helsinki declaration |
| 3. | Has had an ileostomy for more than 3 months | To ensure subjects are recovered from stoma surgery |
| 4. | Has suitable peristomal skin area (assessed by investigator) | To be able to have |
| 5. | Is currently using flat SenSura Mio 1-piece or 2-piece | To ensure that the subjects are used to standard Coloplast adhesive |
| 6. | Has used flat SenSura Mio 1-piece or 2-piece for at least 14 days | To ensure that the subjects are used to standard Coloplast adhesive |
| 7. | Has a stoma size less than 45mm in diameter | To ensure Test product fits around the stoma |

# 6.1.2. Exclusion criteria

| | To be included in this investigation the subject must answer no to the following exclusion criteria | Justification for exclusion criteria: |
|---|---|---|
| 1. | Is currently receiving or have within the past 60 days received radio- and/or chemotherapy (Low doses radio- and/or chemotherapy (Assessed by Principal Investigator) is allowed for indications other than cancer) | The skin undergoes major changes as a consequence of ra-<br>dio- and/or chemotherapy, and therefore it can be more frag-<br>ile to baseplate changes |
| 2. | Is currently receiving or have within the past 30 days received topical steroid treatment in the peristomal skin area, e.g. lotion or spray or systemic steroid (tablet/injection) treatment | Steroid product may interfere with the endpoints by making the peristomal skin thinner and more fragile |
| 3. | Is pregnant or breastfeeding | Even though the ingredients and the recipes are biocompatible, their effect on embryos, foetuses, and infants are unknown |
| 4. | Has dermatological problems in the peristomal area (assessed by investigator) | The skin has to be intact in order to see a potential damage of the skin with simulated/real output |
| 5. | Participates in other clinical investigations. Exception: Participation in other Coloplast sponsored clinical investigations is accepted under the circumstances that the subject has paused the activities in the investigation and are otherwise complying with the inclusion and exclusion criteria of this protocol | Other interventional investigation guidelines/products may interfere with these investigational endpoints |
| 6. | Has any known allergies towards ingredients in the investigational device | To ensure subject safety and integrity of results |

# 6.1.3. Pregnancy and breastfeeding

For female subjects with childbearing potential (they have had at least one period during the last 12 months), a urine pregnancy test will be performed at the inclusion visit, to ensure the subject is not pregnant. The urine pregnancy test will be performed by dip-stick at the trial site. Furthermore, the female subjects should not be breastfeeding, when participating in the clinical investigation.

Besides a negative pregnancy test the women must also use safe contraceptives during the study period (i.e. contraceptive coil, hormone based contraceptives or surgical sterilization). However, in some cases when females older than 50 years but not yet post-menopausal, the investigator may evaluate that it is not reasonable to ask these females to start using safe contraceptives for the duration of the investigation and the investigator can include those female subjects.

If the subject becomes pregnant during the investigation, it is important, that the subject informs the Investigator/Investigator representative immediately. The investigator will then consider whether she should continue in the investigation.

# 6.1.4. Vulnerable population (If applicable)

Not applicable.

### 6.2. Recruitment and enrolment

| Recruitment method | |
|---|---|
| Potential subjects | |
| First contact | |
| Second contact | If potential subjects reply to the email or have called the investigator as first contact and are interested, the Investigator or delegated site personnel will contact the subjects by phone and give a short introduction to the investigation and go over the inclusion and exclusion criteria. If the subjects do not meet the inclusion criteria or meet the exclusion criteria, this will be registered in the Subject Screening Log. |

| Recruitment method | |
|---|---|
| Subject Infor-<br>mation Form | If subjects are eligible and interested in participating, then written information about the investigation (subject information) will be sent to the subjects to ensure that they are given the opportunity to read about the investigation before a possible informational visit, and so that they can prepare any possible questions they may have. Information visit V0 will be booked at this point and the subjects are instructed to contact the investigator or delegated study personnel if they, after having read the subject information, no longer are interested in participation in the study. |
| First visit<br>Information visit | If an eligible subject is interested in participating, information visit (V0) will be arranged in a room ensuring quiet surroundings. That could either be in the subject own home or at Coloplast if preferred by the subject. When arranging the visit, it will be ensured, that the subject has received the Subject Information prior to the visit. The subjects will receive both written and verbal information about the possibility of bringing a companion to the informational visit and to any possible subsequent visits. |
| | for information to be given to the subjects, as well as the informed consent process. |
| Enrolment and in-<br>clusion visit (V1) | The subjects have the right to wait 24h before deciding on participation. If/when the subject decides to participate he/she will be asked to sign the relevant forms (see section 13). If a subject so desires, and it is certain that it is understood what the investigation entails and the relevant forms have been signed the subjects are considered enrolled in the investigation. |

## 6.3. Subject withdrawal criteria

The subject is allowed to withdraw from the investigation at any time for whatever reason without any consequences for their future treatment outside the clinical investigation. The Investigator may withdraw a subject from the investigation at any time if they judge it to be the subject's interest.

The investigator must withdraw a subject from the investigation due to:

- Noncompliance with the CIP impacting the scientific integrity of the investigation.
- If subject's safety and wellbeing is compromised by further participation.
- Subjects lost to follow-up. At least three documented attempts will be made to verify subjects lost to follow-up.

Screening failures and subjects who withdraw or are prematurely terminated from the investigation will be replaced until 10 subjects have completed the study.

A subject who is withdrawn from the investigation, for any reason, will be encouraged to contact the PI if problem arises that the subject believes are related to the clinical investigation. Subject who has not experienced any adverse events, will not be followed up. For subjects who experience adverse events see section 18.1.

### 6.4. Point of enrolment

A subject is considered enrolled in the investigation at the time at which, following recruitment and before any clinical investigation-related procedures are undertaken, the subject signs and dates the informed consent form. The expected duration for each subject is described in section 5.1.

### 6.5. Subject Identification and Confidentiality

Subjects will be identified on the electronic CRF (eCRF) or paper CRF and any other document transmitted to the sponsor by the principal investigator or clinical site staff, by a unique identification number.

Data entered on the eCRF or paper CRF are confidential and will only be available to the sponsor (including sponsor delegates), members of the EC and if requested to regulatory authorities.

The principal investigator for each clinical investigation site will as part of the investigational file maintain a list identifying all subjects entered into the clinical investigation.

### 7. Procedures

# 7.1. Clinical investigation-related procedures

#### Visit 0

Introduction to the investigation

### Visit 1 (It is possible to perform V0 and V1 on the same day)

- Informed Consent Form signed
- Register date of visit
- Allocate subject number
- · Check of inclusion and exclusion criteria, including pregnancy test, if applicable
- Registration of baseline data
  - Age [years]
  - Gender [Male/Female]
  - Height [cm]
  - o Weight [kg]
  - Year of creation of stoma [year]
  - What was the reason for creation of your stoma [Morbus Crohn, Colitis ulcerosa, Cancer, Other (text)]
  - What is your current product size (baseplate size) Length [mm], Width [mm]
  - What type is your current SenSura® Mio product? [1-piece/2-piece]
  - Which stoma accessories do you normally use? (You may tick more than one box) [None/Adhesive remover/Paste/Rings/Stoma tape/Stoma belt/Hernia belt/Stoma powder/(Barrier lotion/cream/spray/wipes)/(Cleansing wipes/cleansing spray)/Odour remover/Other accessories (text)]

Use of accessories are allowed as long as they are not used in the area around the stoma (~3-5 mm) during visits.

### Visit 1-2 (Testing Test product A and B)

- Visual inspection of whether the subject has suitable peristomal skin area for the test (assessed by Investigator, or designee). If the peristomal skin is deemed unsuitable for the test the visit must be rescheduled (if the subject has been rescheduled twice and the peristomal skin is still not deemed suitable for the test the subject will be terminated and replaced)
- Subject questions regarding the perception/condition of their peristomal skin (PIB)
- Measure the diameter of the subject's stoma (done by Investigator, or designee)
  - Diameter of the stoma on the widest place [mm]
  - o Diameter of the stoma on the smallest place [mm]
  - Shape of the stoma [Round/Oval/Irregular]
- Take photos of the peristomal skin before application of the Test product
- Take photos of the Test product when cut to fit the stoma (adhesive site)



Just before removal of the Test product ask the subject to complete questions regarding the perception/condition of their peristomal skin (PIB)

- Assess the subject's wellbeing and compliance with the CP363 clinical investigation plan
- · Assess and record any deviations and adverse events
- Record any given concomitant medication
- Perform device accountability
- Schedule next visit

# Addition to Visit 2 (Testing Test product B) - Termination visit

Fill in the Termination Form

### 7.2. Flow-chart

Table 1 chart showing the connection between visits and assessments.

| | 90000000000000000000000000000000000000 | | | | |
|---|---|---|---|---|---|
| | PER-<br>FORMED<br>BY | SCREEN-<br>ING<br>(V0) | VISIT 1<br>(V1) | VISIT 2<br>(V2) | TERMINA-<br>TION<br>(V2) |
| General | | | | | |
| Oral information | Investigator | х | | | |
| Written informed consent | Investigator | | х | | |
| Check of in- and exclusion criteria | Investigator | х | x | | |
| Insurance of subjects' wellbeing and compli-<br>ance with CIP | Investigator | х | х | х | Х |
| Baseline data | | | | | |
| Registration of baseline data | Investigator | | х | | |
| Registration/measurement of end points | | | | | |
| Visual inspection of whether the subject has suitable peristomal skin area for the test (assessed by Investigator, or designee). If the peristomal skin is deemed unsuitable for the test the visit must be rescheduled (if the subject has been rescheduled twice and the peristomal skin is still not deemed suitable for the test the subject will be terminated and replaced) | Investigator | | X | × | |

| Subject questions regarding the perception/condition of their personal skin (PIB) Measure the diameter of the subject's stornal (done by investigator, or designee) Diameter of the storna on the widest place (mm) Diameter of the storna on the widest place (mm) Diameter of the storna on the smallest place (mm) Diameter of the storna on the smallest place (mm) Shape of the storna (Round/Coval/irregular) Investigator Inv | | | | |
|---|---|---|---|---|
| Measure the diameter of the subject's stormal (done by Investigator) | Subject questions regarding the perception/condition of their peristomal skin (PIB) | Subject | Х | Х |
| Diameter of the stoma on the widest place [mm] Diameter of the stoma on the smallest place [mm] Shape of the stoma [Round/Oval/Irregular] Investigator I | | Investigator | × | Х |
| Investigator X | Diameter of the stoma on the widest place | Investigator | × | Х |
| Investigator | | Investigator | x | Х |
| Investigator | Shape of the stoma [Round/Oval/Irregular] | Investigator | х | Х |
| Investigator | | Investigator | x | Х |
| Investigator | | Investigator | х | Х |
| Investigator | | Investigator | x | Х |
| Investigator | | Investigator | х | Х |
| Investigator | | Investigator | Х | Х |
| Investigator X X X | | Investigator | Х | Х |
| Investigator X X X | | Investigator | Х | Х |
| Investigator X X Investigator | | Investigator | х | Х |
| Investigator X X Investigator | | Investigator | Х | Х |
| Investigator X X X | | Investigator | Х | Х |
| Investigator X X X Investigator X X X X | | Investigator | x | X |
| Investigator X X X Investigator X X X X Investigator X X X X X X X Investigator X X X X X X X X X X X X X X X X X X X | | Investigator | Х | х |
| Investigator X X X | | Investigator | х | x |
| Investigator X X Investigator | | Investigator | Х | Х |
| Investigator X X Investigator | | Investigator | х | Х |
| Investigator X X Investigator | | Investigator | х | х |
| Investigator X X Investigator X X Investigator X X Investigator X X Assess the subject's wellbeing and compliance with the CP363 clinical investigation plan Assess and record any deviations and adverse events Investigator X X Investigator | | Investigator | х | х |
| Investigator X X Investigator X X Assess the subject's wellbeing and compliance with the CP363 clinical investigation plan Assess and record any deviations and adverse events Record any given encomitant medication | | Investigator | х | Х |
| Assess the subject's wellbeing and compliance with the CP363 clinical investigation plan Assess and record any deviations and adverse events Investigator X | | Investigator | х | Х |
| Assess the subject's wellbeing and compliance with the CP363 clinical investigation plan Assess and record any deviations and adverse events Investigator X X X X X X X X X | | Investigator | х | Х |
| ance with the CP363 clinical investigation plan Investigator Investiga | 28次代码。1440年 | Investigator | х | Х |
| Assess and record any deviations and adverse events Investigator X X X | ance with the CP363 clinical investigation | Investigator | х | х |
| Pagerd any given concenitant medication | Assess and record any deviations and ad- | Investigator | х | Х |
| | | Investigator | х | Х |
| Perform device accountability Investigator X X | Perform device accountability | Investigator | х | Х |

| Registration of termination | | | | |
|-----------------------------|--------------|---|---|---|
| AEs/ADEs/SAEs/SADEs | Investigator | х | Х | × |
| Termination form | Investigator | | | × |

## 7.3. Concomitant treatment

Concomitant treatment, including relevant medication, will be registered in the (e)CRF.

There are no restrictions regarding concomitant treatment, besides for those mentioned in the exclusion criteria

# 8. Risk - benefit analysis and ethical considerations

### 8.1. Risk-benefit analysis of the investigational device

A few risks connected to use of the prototypes have been identified in the Product Risk Assessment (9). All risks will be mitigated before release of products for the clinical investigation.

The risk management process has been performed in accordance with the requirements stated in ISO 14971:2012 and in accordance with internal Coloplast procedures, including design verification, validated test methods, risk analysis and completion of a biological evaluation report for the prototypes.

Risks have been proven minimized or eliminated through appropriate design control, confirmed by pre-clinical bench, laboratory and animal testing. The following risks will be mitigated by actions during the clinical investigation.



The investigation is conducted in accordance with current law and applicable standards. Please refer to section 15, Statement of compliance. The rights, safety and well-being of human subjects shall prevail over the interest of science of society.

# 8.2. Risk-benefit for subjects participating in the clinical investigation

The investigation is conducted in accordance with current law and applicable standards, see section 15. Statement of Compliance. The rights, safety and well-being of human subjects shall prevail over the interest of science of society.

Risks in this investigation are considered to be equal to the use of ostomy products already on the market. Risks associated with the use of ostomy products are skin irritation. Please also see Adverse events, adverse device effects and device deficiencies section 18.

There is no known interaction between the use of the Test Product and the medication participants can take – except from what is stated in the exclusion criteria. Disadvantages of testing (trial engagement) may be the time spent on visits.

There are no specific benefits associated with participation in this study other than the participating subjects will contribute with important information for developing new ostomy products.

# 8.3. Risk Analysis for the conduct of the clinical investigation

A risk assessment of the clinical investigation will be conducted initially prior to the first subject enrolment and periodically re-assessed based on any new risks identified through the process. This assessment will be completed throughout the duration of the investigation, as defined by the study team. A risk-based monitoring strategy may be implemented including on-site remote, and central monitoring. Details of the strategy are defined in the monitoring plan.

### 8.4. Delegation of responsibility

Before initiation of the clinical investigation, sponsor must be provided with key personnel signed and dated curriculum vitae (not more than 2 years old) to verify their qualifications. Key site personnel are those, who treat or evaluate subject data in the clinical investigation. Also, the sponsor will ensure that all site personnel are trained in the investigation procedures, how to complete the CRFs, procedure for reporting an adverse event or serious adverse event (how, when, to whom), and who to contact in case of emergency related to the investigational device.

# Monitoring activities

The sponsor is responsible for ensuring appropriate monitoring of the clinical investigation activities as described below.

The monitors will be the primary contact for the principal investigator and clinical investigation site personnel.

Monitoring activities are mandatory as per good clinical practice, however the extend and depth of these activities depend on the criticality of the clinical investigation, speed of enrolment, the experience of the clinical investigation site personnel in carrying out clinical investigations and specific study designs.

## 9.1. Site visits

For the purpose of this clinical investigation the below described monitoring procedures have been determined.

### 9.1.1. Site selection visit

Depending on the prospective clinical investigation sites experience with the specific investigational device, an on-site qualification or site selection visit shall be performed during which the feasibility of the clinical investigation requirements will be discussed and common agreement between sponsor and principal investigator shall be reached. This visit may also be replaced by one or more phone calls if the principal investigator is known to the sponsor.

### 9.1.2. Initiation visit

The clinical investigation site will complete an initiation visit during which full training on all aspects of the clinical investigation will be provided.

### 9.1.3. Monitoring visit(s)

The sponsor shall determine the extent and nature of monitoring appropriate for the clinical investigation based on the risk assessment. The sponsor shall ensure, through oversight of the clinical investigation and timely adverse event reporting, that unanticipated adverse device effects are identified and investigated rapidly so that, where necessary, additional risk control measures can be implemented.

The site dedicated monitor is to ensure adherence to the clinical investigation plan, the safety of the subjects, accurate data recording on the e-CRFs and to monitor recruitment rates and adherence to follow-up schedules. During the clinical investigation, monitors shall check that appropriate written informed consents have been obtained. The principal investigator shall permit and assist the monitor to carry out verification of completed e-CRFs against data in the source documents.

The principal investigator can delegate tasks to his/her collaborators, however the roles and responsibilities as time period of involvement for each clinical site personnel must be documented on the Site Personnel signature and Delegation list as well as training received before getting involved with the clinical investigation must be documented in the Clinical Investigation Training Log.

The monitor shall inform the sponsor about any problems relating to facilities, technical equipment, or site personnel at the clinical investigation site. The monitor shall also be responsible for notifying such deficiencies in writing to the principal investigator and convene with the clinical investigation site personnel appropriate and timely corrective actions.

The sponsor, or delegate, will provide clinical monitoring, including review of eCRF with verification to the source documentation, as defined below or in the monitoring plan.

- At a monitoring visit all available data in the eCRF must be monitored including verification of all fields in the eCRF
- Within 4 weeks after a subject has completed/terminated the investigation, all data should be monitored and all queries related to the subject must be resolved and closed Fourteen days before planned LPO, the monitoring and verification of all available data in the eCRF must be finalised and all available queries must be resolved and closed.
- For subjects terminating the investigation within 14 days before planned LPO, monitoring and verification of data must be finalized within 2 days after the subject's termination visit.
- After LPO, monitoring and verification of data must be finalized within two days after LPO.
- Queries raised after LPO must be resolved within two days.
- At the Monitoring Visits before the planned LPO, the monitor must ensure PI readiness for signing the eCRF (has completed relevant eLearning in the eCRF) and is available for signature after LPO. In addition, ensure site personnel is available for query resolution after LPO, if raised.

The monitor shall make written reports to the sponsor, including documentation of any deviations after each visit and provide written follow up action items if any, to the principal investigator and/or clinical investigation site personnel.

Source data verification will be performed to the extent it is possible. The Source Data Specification Form must be completed at the initiation visit detailing the location of the source data for each data point. Where no source data (besides the eCRF) is available the contents of the eCRF will be monitored.

The Informed Consent Forms and AE/ADE will be 100% monitored for timely completeness.

Only the investigator, delegated site personnel and the sponsor representatives will have access to all the eCRFs.

### 9.2. Remote monitoring

Remote (source data verification) and/or centralized (data review) monitoring is carried out by sponsor personnel or representatives (e.g., data management personnel, statisticians, or clinical monitors) at a location other than the site(s) at which the clinical investigation is being conducted (evaluation without visiting the investigation site). Remote monitoring processes can provide many of the capabilities of on-site monitoring as well as additional capabilities.

In addition to onsite monitoring visits, remote monitoring of the data entered in the e-CRF system could be used to achieve the following:

- Conduct activities such as: standard checks of range, consistency, and completeness of data and checks for unusual distribution of data, such as too little variance)
- Special attention will be given in case of frequent data anomalies or errors, protocol deviations or excessive dropouts.

- Augment on-site monitoring by performing monitoring activities that can only be accomplished using centralized processes
- Monitor data quality through routine review of submitted data in real-time to identify missing data, inconsistent data, data outliers, and potential protocol deviations that may be indicative of systemic and/or significant errors in data collection and reporting at the site
- Verify source data remotely, provided that both source data and CRFs can be accessed remotely
- Conduct analyses of site characteristics, performance metrics (e.g., high screen failure rates, high
  frequency of eligibility deviations, and delays in reporting data), and clinical data to identify early on
  corrective actions needed for characteristics correlated with poor performance or noncompliance

### 9.3. Source data verification

Source data is all information in original records, certified copies of original records of clinical findings, observations, or other activities in the clinical investigation, necessary for the reconstruction and evaluation of the clinical investigation. This includes source data initially recorded in an electronic format.

All documents and data related to the clinical investigation handled by site personnel, shall be produced and maintained in a way that assures reliability, integrity, control and traceability, and shall be appropriately stored to provide a complete history.

The Principal Investigator shall assure the accuracy, attribution, completeness, legibility and timeliness of the data reported to the sponsor in the eCRFs and in all required reports. All printed copies of electronic source documents shall be certified, as indicated by a dated signature by the investigational site personnel at the time the document is printed. Special requirements should be applied to the capture, review and retention of electronic source data, to ensure reliability, quality, integrity and traceability.

The data reported in the eCRFs shall be derived from source documents and be consistent with these source documents, and any discrepancies shall be explained in writing. The eCRF can serve as the source document and this must be documented on the Source Data Specification Form. The Source Data Specification Form must be completed at the initiation visit detailing the location of the source data for each data point agreed upon by the Principal investigator.

### 10. Statistical considerations

# 10.1. Statistical design, method and analytical procedures

# Definition of analysis populations

Intention to Treat (ITT) and Safety populations will be defined at a formal data review meeting before data-base lock. As a minimum, the data manager, the clinical manager and the statistician will be involved in the classification of subjects.

The ITT population (full analysis set) will be constituted by all subjects with valid informed consent who have been exposed to at least one Test product, with information on at least one endpoint.

The Safety population will constitute by subjects who have given informed consent.

All evaluations of endpoints will be based upon the ITT population whereas adverse events will be assessed based on the safety population. Invalid individual data points may be omitted from evaluations even though the corresponding subject is part of the ITT population. Any exclusion of data points will be documented.

Considering the data obtained it might be considered to make additional explorative analyses based on a subset of the ITT population.

Evaluation of endpoints and individual questions

All endpoints and individual questions from questionnaires will be listed and summarized by descriptive statistics. The summaries and listings will be done by Test product. For relevant questions, the summaries will be done before and after use of the Test products.

Summary statistics for continuous variables are presented with N, Mean, SD (standard deviation), Median, Min and Max, where N denotes the number of subjects contributing with non-missing data. For discrete variables, summary statistics are presented with N and percentage, where percentage is based on the total number of subjects/observations with non-missing data.

The PIB score is calculated as the maximum value of the 3 individual measures of Pain (0-10), Itching (0-10) and Burning (0-10).

Other summaries and analyses can be made, if relevant.

All statistical summaries and listings are made with SAS version 9.4 (SAS Institute Inc., Cary, NC)

### 10.2. Sample size

As this is an exploratory investigation with a qualitative primary outcome no formal sample size is calculated but it is evaluated that 10 subjects with an ileostomy (liquid output) will be adequate to investigate Test product A and B's ability to swell around the stoma.

# 10.3. Level of significance and power

The data will primarily be evaluated based on summary statistics. If explorative statistical analyses are performed a significance level of 5% will be applied.

#### 10.4. Pass/fail criteria

This is an exploratory investigation and there is no formal success and/or fail criteria.

### 10.5. Interim analysis

There is no planned interim analysis in this investigation.

# 10.6. Statistical reason for termination of investigation

There will be no interim analysis and therefore no reason to terminate the investigation based on statistical considerations.

# 10.7. Deviation(s) from statistical design, method or analytical procedures

Any deviations from the statistical plan will be documented in the clinical investigation report.

# 11. Data management

Data management of all measurements described in this protocol are carried out by Clinical Operations, Coloplast A/S.

Data will be collected through an electronic data capturing (EDC) system on electronic Case Report Form (eCRF), a secure, internet-based case report form.

The EDC system used is

The system is designed to be compliant with the FDA requirements of 21 CFR part 11. It is a validated data management system, with restricted role-based access control, allowing only qualified and trained personnel to enter the system. The system has full audit trail and electronic signature.

The principal investigator and delegate(s), and investigation monitor(s) must be trained in the system prior to getting access. The training is web-based (eLearning) and must be completed before access to the investigation is granted. The web-based training will be documented in the data management system. In addition, the data management specialist will demonstrate the system on a virtual/physical meeting. This training will be documented in the Clinical Investigation Training Log. The sponsor will be responsible for training the investigator, delegate(s) and the monitor(s).

Only the principal investigator, or delegate(s), who have completed the relevant eLearning, signed the Site Personnel Signature and Delegation List and Clinical Investigation Training Log will be authorised to enter data in the eCRF. When training is completed site personnel will initially get access to a training/sandbox database, for the site to get access to the real database as a minimum the Principal Investigator at a site the must complete.

The eCRF will be completed by the investigator, or delegate, that will perform primary data collection directly into the eCRF or drawn from source-documents and by the subject. The eCRF will be completed on a continuous basis starting from the point of enrolling the subject to final follow up. In addition, the principal investigator, using his/her personal login information, will be authorised to, and must, sign each eCRF. It will also be the responsibility of the investigator to ensure that all measurements and observations are correctly noted in the eCRF.

The investigator will keep a separate list of the subjects' ID numbers, names, and addresses in a locked room/cabinet.

The monitor, using his/her personal login information shall verify all data points and issue electronic queries for the authorised clinical site personnel to respond, as defined in the monitoring section (and monitoring plan, if created).

The Data Validation Plan describes which edit checks, range checks, and other consistence checks that will be done on the clinical data during conduct of the investigation. The Data Validation Plan will be developed in collaboration with the Clinical Manager and the Statistician and will be aligned with the monitoring section (and monitoring plan, if created).

A critical quality control will be performed by the data management team and queries issued where needed. Such queries must be resolved by the site personnel. Automated, real-time access to the data enable control on study compliance and safety assessments. A full audit trail ensures, that each user's (site personnel, monitor, sponsor, data manager) access to and actions in the system is tracked.

At the end of the study formal data review meeting(s) will be performed before the database will be locked.

The Data Management procedures are further described in the Data Management instructions.

### 11.1. Data collection procedure

All assessments and observations throughout the investigation for each subject must be carefully recorded in an eCRF or in a paper CRF (pCRF) during the visit or immediately after. The eCRF makes it possible to enter data right away when they are obtained. This is the preferred way of collecting data. In case this is not possible the data should be entered no later than seven days after the visit / procedure.

When subject and investigator is required to complete different sections in the CRF, it will be specified which sections the subject will fill in (using paper CRF or app solution) and which sections the investigator will fill in.

In the unforeseen situation, where site cannot establish connection to the EDC system, a paper CRF (pCRF) has been printed and supplied by sponsor.

If for some reason is not available the subject must complete the questionnaire on the paper CRF, and the data must be entered into the eCRF by site personnel.

Qualitative evaluations will be registered in an Excel Sheet, that will be saved in the Data Management archive site with data management access only. Only the overall conclusions will be registered in the eCRF.

Photos and video records will be saved in the Data Management archive site with data management access only.

The remaining endpoints, assessment, backup measurements and baseline information can be entered directly into the eCRF.

### 11.2. Data retention

The Investigator file must be archived for a minimum period of 10 years after the final clinical investigation report has been signed.

# 12. Amendments to the Clinical Investigation Plan

No changes in the clinical investigation procedures shall be affected without mutual agreement between the principal investigator and the sponsor. The agreement of the changes must be documented by signing the corresponding clinical investigation plan amendments and registered in the Change Log.

All significant changes require notification to the EC and applicable regulatory authority. Substantial changes may require approval from the EC and applicable regulatory authority prior to implementation. (Example of significant change: Changes of inclusion criteria, end points or assessment methods)

# 13. Deviations from the Clinical Investigation Plan

Deviations to the Clinical Investigation Plan occurs when the activities during the clinical investigation do not comply with the EC approved investigation plan.

The investigator is not allowed to deviate from the Clinical Investigation Plan unless, under emergency circumstances or to protect the rights, safety and welfare of the subject(s).

If a situation occurs, that affect the rights, safety and well-being of the subject(s), the investigator is obliged to deviate from the CIP, and other regulations to protect the subject. The Investigator must inform the monitor immediately, and the Monitor will report and inform the Clinical Manager or designee immediately. Documentation with all relevant details will be completed to document the deviation and must be reported to the EC by the CM as required by local regulations.

The site will complete a protocol deviation eCRF form for all subject-related deviations and all deviations that are <u>not</u> related to a subject (for example, an untrained nurse performing study procedures) are reported in the Deviation Log by the investigator.

If any deviations to the investigation plan are detected during the monitoring visit, the Monitor shall ensure the site reports all subject-related deviations in the eCRF and non-subject related deviations on the Deviation log in the Investigator File. Additionally, the monitor must report any deviation noted during the visit in the Periodic Monitoring Report.

### 14. Device Accountability

All access to the investigational devices used in the clinical investigation is controlled by storage procedures and device accountability logs as described below. The investigational devices must only be used in this clinical investigation and only according to the CIP.

Sponsor keeps a device accountability log that states the physical location of all investigational devices from shipment of investigations devices to the investigational sites until return of or disposal.

The PI or an authorized designee keeps records documenting the receipt, use and return and disposal of the investigational devices, which includes:

- Date of receipt.
- Identification of each investigational device (batch no./serial no./unique code).
- The date(s) of use.
- · Subject identification.

### 15. Statement of compliance

The clinical investigation is conducted in accordance with:

- Ethical principles that have their origin in the Declaration of Helsinki, 1964, Last amended at the 59th WMA General Assembly, Brazil, October 2013.
- MDR (EU) 2017/745
- ISO 14155:2020 "Clinical Investigation of medical devices for human subjects Good clinical practices".
- Any applicable regional or national regulations will be specified in the country specific CIP.

### 15.1. Ethics committee and regulatory authorities

The CIP and/or other relevant documents are submitted to the appropriate EC(s). This clinical investigation will not begin until the required approval from the EC has been obtained. Any amendment to the protocol will be submitted to the same EC(s).

Sponsor will notify the EC(s) concerned of the end of the clinical investigation.

### 15.2. Data protection

As part of the investigation Coloplast A/S, ("Coloplast") will collect and process the personal information the subject provides for the investigation ("subject personal data"). This includes identification and contact information (which may be anonymised depending on the nature of the investigation) as well as information about product usage experience and your health. Coloplast will comply with the EU General Data Protection Regulation (GDPR) and the Danish act on data protection ("databeskyttelsesloven"), including in connection with transfer of data to third countries, cf. chapter V of GDPR, Coloplast will only process the subjects' personal data:

- 1. To conduct the investigation and carry out related research based on subject consent (primary use), cf. articles 6(1)(a) and 9(2)(a) of GDPR,
- 2. To comply with applicable legal obligations to e.g. ensure reliability and safety, cf. article 6(1)(c) in conjunction with article 9(1)(i) of GDPR, and
- 3. If separate consent is given for secondary use of subject personal data, cf. articles 6(1)(a) and 9(2)(a) of GDPR carry out research outside the clinical protocol to improve Coloplast's products and services, and for use in education.

Part of Coloplast's processing is carried out on third-party platforms (clinical trial databases) and certain third parties are assisting Coloplast in the processing (e.g. the investigator). Such cases will imply a transfer of your personal data to the third parties, but solely for the specified purposes and with the third parties acting on

instruction from Coloplast. Data may be collected and processed across the Coloplast network, which may entail processing of personal data outside the European Economic Area. In such cases, an adequate level of protection will be ensured by the third parties being subject to the standard contractual clauses on data protection adopted by the EU or to an EU-approved certification mechanism on data protection. For further information about this please the subject can always consult Coloplast's data protection officer (details below).

Subject personal data will be kept as long as required under applicable laws and regulations. The EU Medical Device Regulation obligates Coloplast to keep the data for a period of at least ten years after the investigation is completed, or, in the event that the device is subsequently placed on the market, at least ten years after the last device has been placed on the market. Subject personal data will be deleted at the end of the mandatory retention period.

If the subject has questions or queries regarding Coloplast's handling of personal information, the subject can always contact Coloplast's Data Protection Officer at Complaints related to Coloplast's handling of subject personal information may similarly be sent to the Data Protection Officer, and the subject is also entitled to file a complaint with the relevant supervisory authority, which in the case of Denmark is the Danish Data Protection Agency (<a href="www.datatilsynet.dk">www.datatilsynet.dk</a>).

The subject can write to

at any time to request:

- Access to personal data
- Correction of errors in personal data or to erase personal data
- Limit what can be done with personal data
- To receive personal data in machine-readable format (data portability).
- Withdrawal of consents the subject has given Coloplast to process personal data

### 15.3. Indemnity

All subjects are fully covered by Coloplast A/S insurance throughout the investigation.



### 15.4. Financial conditions

Coloplast A/S will compensate all investigators involved in the clinical investigation for their time and resources spent on the investigation. All financial agreements with the investigation sites involved in the clinical investigation will be specified in a sponsor investigator agreement.

The budget includes the salary to the Principal Investigator and study nurses, the cost of Test Products, transportation, and gift vouchers to the subjects. The Principal Investigator and study nurses have no financial interest in the investigation. The total budget for the investigation is covering 10 participants.

# 16. Informed consent process

Written informed consent is obtained from all subjects participating in the investigation after thorough written and verbal information. The information is given by the investigator or his/her representative in the subjects' native non-technical language. Each subject will be fully informed about the aim of the investigation, procedures, potential risks or inconveniences and/or expected benefits, all anticipated adverse device effects and then have a minimum of 24h before deciding on participation. The subjects will be informed that their participation is voluntary and that they may leave the investigation at any time, without this having any influence on their further treatment.

The informed consent signature form includes personally dated signatures of the subject and the PI or his/her representative responsible for conducting the informed consent process. A copy will be provided to the subject.

If new information is to be given during the investigation, sponsor will inform the investigators, and the new information is given to the subjects by the investigator. If new information becomes available that can significantly affect a subject's future health and medical care that information will be provided to the subject in written form. CM is responsible for writing the information and providing the approved Subject Information and Consent Form to investigators that will further provide it to the subjects. If applicable, all affected subjects shall be asked to confirm their continuing informed consent in writing.

This procedure also applies to informed consent obtained from a subject's legal representative. The procedure cannot waive the subjects' legal rights.

# 17. Subject compensation

### 17.1. Compensation in case of injury

Product liability and No-Fault Clinical Investigation Insurance covering the duration of the clinical investigation are in place, to enable compensation in the event of an injury to a participating subject. See section 15.3.

# 17.2. Compensation for participating in the clinical investigation

Transport between Coloplast and Subjects home will be covered. Reimbursement of transport expenses are not taxable Transport expenses will be paid in appropriate portions that justify the administration, throughout investigation period.

# 18. Adverse events, adverse device effects and device deficiencies

#### 18.1. Adverse events

An adverse event is any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, whether or not related to the investigational medical device(s) or the comparator(s), or the procedures involved. The adverse event shall be marked with the intensity mild, moderate or severe. This could include events such as headache or dizziness.

### 18.2. Adverse device effect

An adverse event, which is related to the use of the investigational medical device, is an adverse device effect, and should be marked as unlikely related, possible related, probable related or with causal relationship on the adverse event form.

The definition of an adverse device effect includes any event resulting from insufficiencies or inadequacies in the instruction for use or any malfunction of the medical device, as well as any event resulting from use error or from intentional misuse of the device.

Table 2 lists anticipated adverse device effects that may occur.

Table 2 Anticipated adverse device effects and their likely incidence rates

| ANTICIPATED ADE | INCIDENCE RATE |
|---|---|
| Peristomal skin irritation (incl. mechanical trauma and skin maceration) | < 10% |
| Allergic peristomal skin irritation (dermatitis) | < 1% |

Temporary redness upon removal of the base plate is not considered an adverse device effect, however an abnormal development in intensity or duration should be considered as such.

### 18.3. Device deficiency

A device deficiency is the inadequacy of the investigational medical device or comparator with respect to its identity, quality, durability, reliability, usability, safety or performance. This includes malfunctions, use errors and inadequacy in the information supplied by the manufacturer including labelling.

Example: Inadequate welding of test product.

#### 18.4. Serious adverse events (SAE)

A serious adverse event is an adverse event that:

- · Led to death.
- Led to a serious deterioration in the health of the subject, users or other persons as defined by one or more of the following:
  - 1) a life-threatening illness or injury, or
  - 2) a permanent impairment of a body structure or a body function including chronic diseases, or
  - 3) in-patient or prolonged hospitalization, or
  - 4) medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function.
- Led to foetal distress, foetal death, a congenital abnormality or birth defect including physical or mental impairment.

This includes device deficiencies that might have led to a serious adverse event if:

- 1) Suitable action had not been taken, or
- 2) Intervention had not been made, or
- 3) Circumstances had been less fortunate.

These are handled under the serious adverse event reporting.

Planned hospitalization for a pre-existing condition, or a procedure required by the CIP, without serious deterioration in health, is not considered a serious adverse event.

### 18.4.1. Serious adverse device effect (SADE)

A serious adverse device effect is an adverse device effect that has resulted in any of the consequences characteristic of a serious adverse event.

### 18.4.2. Anticipated serious adverse device effect (ASADE)

Anticipated serious adverse device effect is any event that by its nature, incidence, severity, or outcome has been previously identified in the risk analysis report. In this investigation no SADE are anticipated.

# 18.4.3. Unanticipated serious adverse device effect (USADE)

An unanticipated serious adverse device effect is a serious adverse device effect which by its nature, incidence, severity or outcome has not been identified in the current version of the risk analysis report.

#### 18.5. Medical care of subjects

Principal investigator shall ensure that adequate medical care is provided, during and after participation in the clinical investigation, to a subject experiencing an adverse event. All ongoing ADEs, SAEs, SADEs and DDs that could have led to a SAE at subject termination will be followed according to the Risk Benefit analysis (see 8.2) and will be followed until a resolution is addressed for a period of 2 months after subject termination. An ongoing adverse event at subject termination visit is documented as the current status for the adverse event and will not be followed up.

The subjects shall be informed of any new significant findings occurring during the clinical investigation, including the need for additional medical care that can be required, and of the nature and possible cause of any adverse events experienced.

### 18.6. Reporting and timelines

## 18.7. Investigator's reporting responsibilities

- Pl at each site must assess all (S)AE's that occur at his/her site.
- All serious adverse events and serious adverse device effects must be reported to sponsor within 24 hours of the site becoming aware of the event.
- A device deficiency that could have led to a serious adverse event but did not because suitable action
  was taken, intervention had been made or because of fortunate circumstances should be reported to
  sponsor within 24 hours of the site becoming aware of the event.
- New findings and/or updates in relation to already reported serious events should also be reported to sponsor within 24 hours of the site becoming aware of the event.

When reporting the SAE, the relationship to the test material shall be described whether the event is considered

- Not related, the event has no temporal relationship with the use of the test material or the procedures.
- Unlikely related, the relationship with the use of the test material seems not relevant and/or the event can be reasonably explained by another cause, but additional information may be obtained.
- Possible related, the relationship with the use of the test material is weak but cannot be ruled out completely. Alternative causes are also possible (e.g. an underlying or concurrent illness/ clinical condition or/and an effect of another device, drug or treatment). Cases were relatedness cannot be assessed or no information has been obtained should also be classified as possible.
- Probable related, the relationship with the use of the test material seems relevant and/or the event cannot reasonably be explained by another cause, but additional information may be obtained.
- Definitely related/Causal relationship, the event has a temporal relationship with the test material use/application or procedures.

and the intensity of the event should be considered, as such:

- o Mild, the intensity of the event is mild with no further action or intervention
- o Moderate, the intensity of the event will lead to an action or intervention to solve the event
- Severe, the intensity of the event will lead to follow up on the action or intervention, as the effect of the action or intervention may not decrease the symptoms.

All above events must be reported by use of the relevant adverse event/serious adverse event/device deficiency form.

### Please report to:



### 18.8. Sponsors reporting responsibilities

It is the responsibility of sponsor to ensure that the following are reported to EC immediately, but no later than 7 calendar days following the date of awareness by sponsor.

- · All serious adverse events.
- All serious device effects.
- All device deficiencies that could have led to serious adverse events but did not because suitable action
  was taken, intervention had been made or because of fortunate circumstances.
- New findings and/or updates in relation to already reported events.

If the serious adverse event results in imminent risk of death, serious injury, or serious illness that requires prompt remedial action for other subjects, users or other persons or a new finding to such a serious adverse event, sponsor must immediately but no later than 2 calendar days after awareness by sponsor report the event to EC.

# 19. Suspension or premature termination of the clinical investigation

Sponsor may suspend or prematurely terminate an investigation site or the entire clinical investigation for documented significant reasons.

If a suspicion of an unacceptable risk to subjects develops during the clinical investigation, sponsor will suspend the investigation while the risk is assessed. Sponsor will terminate the investigation if an unacceptable risk is confirmed. Sponsor will ensure that the premature termination will be justified in writing and will promptly inform the regulatory authorities and relevant EC(s). If monitoring or auditing of the clinical investigation identifies serious or repeated deviations at one of the participating investigation sites, sponsor will suspend or terminate the particular investigational site. The sponsor or investigator will inform the regulatory authority as appropriate and notify the EC about the termination of the site.

If suspension or termination of the clinical investigation occurs, the investigator(s) will promptly inform the enrolled subjects. Sponsor will provide resources to fulfil the obligations from the CIP for follow-up on the subjects as necessary

### 20. Clinical investigation report

At completion of the investigation sponsor is responsible for writing the clinical investigation report. The report is retained on file. The report contains a critical evaluation of all data, which have been collected during the investigation. The report describes the methodology and design and a data analysis, including statistical preparation and conclusion.

Sponsor and investigator must sign the final version of the clinical investigation report or an affidavit, indicating their agreement with the contents. If no coordinating investigator is appointed, then the signatures of the principal investigator(s) should be obtained.

The clinical investigation report must be submitted to EC.

### 21. Publication policy

If the Trial Site, PI and/or the staff involved in the Investigation wish to publish their results of the Investigation, the publication will be sent to Sponsor for prior review no later than thirty (30) calendar days before submitting the publication to the media concerned.

Publication policy is specified in Sponsor Investigator Agreement.

### 21.1. General

The investigation will be registered on a public accessible database, e.g. www.ClinicalTrial.gov, before recruitment of the first subject. The results of the investigation, positive as well as negative, may be communicated

by abstracts, posters or oral presentations provided that opportunity is given for sponsor to discuss the contents and any conclusions drawn, before the abstract, paper or visual presentations are finalised. In all cases the subject's identity will remain confidential.

Sponsor will undertake to comment on the draft documents within 30 working days of receipt, but the final decision on the contents and format of the publication from the conclusions drawn, will remain with the authors.

No preliminary results will be published.

Data from the investigation is considered confidential until it is published according to the conditions of this CIP.

Sponsor may publish single subject case stories at any time during and after the investigation.

Sponsor reserves the right to use the data (published and unpublished) for reimbursement or regulatory purposes.

# 22. Suspension/termination of the clinical investigation

Sponsor will withdraw from sponsorship of the clinical investigation if

- major non-adherence to the clinical investigation plan is occurring.
- it is anticipated that the subject recruitment will not be adequate to meet the investigation objectives [at least 75%] of the subjects should be entered within the recruitment time.

In case sponsor withdraws, sponsorship for the subjects already recruited into the clinical investigation will continue.

# 23. References

- Fellows J, Voegeli D, Håkan-Bloch J, Herschend NO, Størling Z. Multinational survey on living with an ostomy: prevalence and impact of peristomal skin complications. British Journal of Nursing. 2021;30(16):S22-S30.
- 2. Martins L, Samai O, Fernández A, Urquhart M, Hansen AS. Maintaining healthy skin around an ostomy: peristomal skin disorders and self-assessment. Gastrointestinal Nursing. 2011;9(Sup2):9-13.
- 3. Voegeli D, Karlsmark T, Eddes EH, Hansen HD, Zeeberg R, Håkan-Bloch J, et al. Factors influencing the incidence of peristomal skin complications: evidence from a multinational survey on living with a stoma. Gastrointestinal Nursing. 2020;18(Sup4):S31-S8.
- 4. Andersen PH, Bucher AP, Saeed I, Lee PC, Davis JA, Maibach HI. Faecal enzymes: in vivo human skin irritation. Contact Dermatitis. 1994;30(3):152-8.
- 5. Baker M, Greening L. Practical management to reduce and treat complications of high-output stomas. Gastrointestinal nursing. 2009;7(6):10-7.
- 6. Hyland J. The basics of ostomies. Gastroenterol Nurs. 2002;25(6):241-4; quiz 4-5.
- 7. Herlufsen P, Olsen AG, Carlsen B, Nybaek H, Karlsmark T, Laursen TN, et al. Study of peristomal skin disorders in patients with permanent stomas. Br J Nurs. 2006;15(16):854-62.
- Investigators Brochure
- 9.

# 24. Appendix

# Case Report Form – Subject – CP363

| | sit: | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject ID | : | | | | | | | | | |
| (from the st | g questions o<br>oma site to ti<br>eriod slnce y | he edge | of the st | in comp<br>oma ba | g adhes | ive). Pled | ise ansv | around<br>ver each | d your st<br>questio | toma<br>on thinking |
| | L. Please rate<br>e you last cho | | | | | | around | your sto | oma has | been <u>at it</u> |
| 0<br>No itch | 1<br>Very mild<br>itch | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10<br>Worst<br>possible<br>peristom<br>skin itæl |
| worst since | Please rate | inged yo | ale from<br>ur produ | ict (tick | one box | ul the sk<br>only) | | T === | | |
| | | 2 | 3 | | 5 | 6 | 7 | 8 | 9 | 10 |
| 0<br>No pain | Very mild<br>pain | | 3 | | | | | • | | Worst<br>possible<br>peristom<br>skin pai |
| | Please rate since you las | | | | | | | ne skin d | around y | our storno |
| at its worst : | | | | | | | | | | |
| at its worst | | 2 | 3 | 4 | 5 | 6 | | 8 | 9 | 10<br>Worst |

# Signature Page for

| Reason for signing: Approved | Name: Role: Author Date of signature: 19-Dec-2023 11:02:25 GMT+0000 |
|---|---|
| Reason for signing: Approved | Name: Role: Approver Date of signature: 19-Dec-2023 11:07:56 GMT+0000 |
| Reason for signing: Approved | Name:<br>Role: Approver<br>Date of signature: 19-Dec-2023 11:17:42<br>GMT+0000 |
| Reason for signing: Approved | Name: Role: Approver Date of signature: 19-Dec-2023 11:26:58 GMT+0000 |
| Reason for signing: Approved | Name: Role: Approver Date of signature: 19-Dec-2023 11:55:05 GMT+0000 |

Signature Page for